CLINICAL TRIAL: NCT01103622
Title: An Open-label, Randomised, Placebo Controlled, Two-Way Crossover, Phase I Single Centre Study in Type 2 Diabetes Mellitus Patients Treated With Metformin to Evaluate the Pharmacokinetics of Digoxin During Co-administration With AZD1656
Brief Title: Investigate the Effect of AZD1656 on the Pharmacokinetics of Digoxin in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00031
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Type 2; Digoxin; drug-drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — AZD1656; Digoxin

ARMS (2):
- 1 (Experimental): twice daily Day 1 to Day 7; digoxin on day 4
  Interventions: Drug: AZD1656; Drug: Digoxin
- 2 (Placebo Comparator): twice daily Day 1 to Day 7; digoxin on day 4.
  Interventions: Drug: Digoxin; Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Oral tablet bd, step-wise increased dosage
  Arms: 1
Drug: Digoxin — Oral tablet od on Day 4
  Other Names: Digacin
Drug: Placebo — Oral tablet bd, step-wise increased dosage
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether AZD1656 will affect the pharmacokinetics (PK) of digoxin in type 2 diabetes mellitus (T2DM) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed type 2 diabetes for at least 1 year and treated with metformin as a single treatment or in combination with one other oral anti diabetic for at least 2 months prior to screening.
* Body mass index between ≥19 and ≤42 kg/m2.
* Haemoglobin (Hb) A1c ≥6.5% and ≤9.5% at enrolment.

Exclusion Criteria:

* History of cardiovascular disease, eg, left ventricular hypertrophy, uncontrolled hypertension, paroxysmal or persistent cardiac arrhythmia or ischemic heart disease.
* Systolic blood pressure >160 mmHg or diastolic blood pressure >95 mmHg at screening
* Use of amiodarone within 3 months prior to screening and the use of potent CYP450 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
evaluate the pharmacokinetics of digoxin after a single dose when administered alone and in combination with AZD1656 at steady state, by assessment of AUC and Cmax of digoxin | Serial PK blood samples will be taken on days 4-8 during the treatment periods

SECONDARY OUTCOMES:
evaluate the safety of AZD1656 in combination with digoxin by assessment of electrocardiogram, weight, pulse, blood pressure, laboratory variables (including 7-point glucose), physical examination and adverse events. | Safety assessments will be monitored throughout the study, from screening visit until follow up visit.
describe the pharmacokinetics of AZD1656 and its metabolite during concomitant digoxin administration by assessment of AUC(0-24), Cmax, Ctrough, tmax, t1/2 and CL/F (AZD1656 only). | Serial PK blood samples will be taken on days 4-8 during the treatment periods
describe the pharmacokinetics of digoxin when administered alone or in combination with AZD1656 by assessment of tmax and t1/2. | Serial PK blood samples will be taken on days 4-8 during the treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Stanko Skrtic, Study Director — AstraZeneca; Christoph Kapitza, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH; Mirjana Kujacic, Study Chair — AstraZeneca
Locations (1):
- Research Site, Chula Vista, California, United States